CLINICAL TRIAL: NCT03702595
Title: Effects of a Stretching Protocol of Hip Flexors in Patients With Mild to Moderate Hip Osteoarthritis
Brief Title: Effects of a Stretching Protocol in Patients With Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: University of Valladolid (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Principal Investigator, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1955
Record Dates: First submitted 2018-08-17; First posted 2018-10-11 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis; Manual therapy; physiotherapy
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Hip flexors stretching protocol
  Interventions: Other: Hip flexors stretching protocol

INTERVENTIONS:
Other: Hip flexors stretching protocol — Stretching protocol of rectus femoris, vastus lateralis and iliopsoas according to Kaltenborn- Evjenth Orthopaedic Manual Therapy Concept (OMT)

SUMMARY:
Hip osteoarthritis (OA) is one of the most prevalent chronic disease in the world. Clinical guidelines recommend non-pharmacological conservative treatments for the management of OA. Hip flexors seems to play an important role in the development of hip OA but there is no published studies evaluating the results of a stretching protocol of hip flexors in hip OA patients.

The objective of this trial is to evaluate if a stretching protocol of hip flexors is more effective in symptoms, functional capacity , range of motion, strength, muscular length, pain threshold and anxiety and depression compared to control.

For this purpose the investigators conduct a single-group, pretest-posttest clinical trial.The investigators included patients diagnosed of hip osteoarthritis Grade I-III by Scale of Kellgren and Lawrence.

The variables are measured at the beginning and at the end of treatment of the control phase, and at the end of the stretching protocol phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with a X-Ray test
* American College of Rheumatology Criteria

Exclusion Criteria:

* Secondary osteoarthritis by a traumatism, Paget disease, inflammatory or metabolic disease, congenital diseases etc.
* Vascular or neurological disease.
* Musculoskeletal pathologies in lumbar spine, pelvis or lower limbs
* Grade IV in Kellgren and Laurence Scale

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pain intensity | 3 weeks
  Visual Analogic Scale

SECONDARY OUTCOMES:
Functional Capacity | 3 weeks
  The investigators measure the functional capacity with Timed Up and Go test (TUG)
WOMAC questionnaire | 3 weeks
  WOMAC questionnaire
Hip Range of Motion | 3 weeks
  Digital inclinometer according to Pua et al., 2008
Muscular strength | 3 weeks
  The investigators measure the hip strength with a hand held dynamometer (Lafayette)
Muscular length | 3 weeks
  The investigators measure the muscular length with an inclinometer
Pressure Pain threshold | 3 weeks
  Pressure algometry measured by digital algometer
Anxiety and Depression | 3 weeks
  Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Sandra Jiménez del Barrio, Soria
  - Luis Ceballos Laita, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The patient data were confidential and were assigned a number to each patient to maintain confidentiality